CLINICAL TRIAL: NCT00339352
Title: A Family Study of Adults With Glioma
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 999999013; OH99-C-N013
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Glioma
Keywords: Brain; Exposures; Genetics; Glioma; Occupations
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 1: Cases
- 2: Controls
- 3: first-degree relatives of cases/controls

SUMMARY:
To advance understanding of environmental, behavioral and genetic causes of brain tumors in adults, DCEG investigators initiated a multicenter case-control study of malignant and benign tumors in adults in 1994. This four-year study was conducted at participating hospitals in Boston, Phoenix, and Pittsburgh. Eligible cases were individuals greater than or equal to 18 years newly diagnosed with an intracranial glioma, meningioma or acoustic neuroma and treated at one of the participating hospitals. The controls were patients admitted to neurological, neurosurgical or general surgical services at the same three hospitals for any of a variety of non-neoplastic conditions. By the end of the study, 811 brain tumor cases had been accrued.

Information about a broad range of possible environmental, lifestyle, and genetic risk factors was obtained from both cases and controls through a computer-assisted personal interview (CAPI). The family history component obtained history and age at diagnosis of cancer or benign brain tumors and selected other diseases, for all living and deceased first degree relatives. A supplemental self-administered questionnaire covered diet, vitamin supplements, alcohol consumption, and household use of electrical appliances. Blood samples were obtained as a source of DNA. Currently, data analysis is in the early stages.

To increase our ability to examine both genetic and environmental components of brain tumor risk, we decided to add a family studies component to the case-control study, focusing on families of glioma cases. Initial contact with each family is made through the cases or, if a case is deceased, through the next of kin. Cases or next of kin are asked to complete a Family Health Questionnaire that updates the family medical history and provides contacting information for all adult first degree relatives and more distant relatives with cancer. Then, we contact all first degree relatives greater than or equal to age 18 years, and the next of kin of deceased eligible relatives and invite them to complete a modified risk factor interview conducted over the telephone. This interview obtains information about each relative s personal and family history of cancer and other diseases, and history of risk factor exposures, including all the major categories covered in the case-control study. Study participants who complete the interview are then asked to provide buccal cells as a source of DNA for future genotyping.

The glioma cases and their relatives will serve as a unique resource for both epidemiologic and genetic analyses. Selected relatives can serve as controls for association thereby eliminating concerns and population stratification. The study design also permits assessment of specific genetic hypotheses that cannot be evaluated in a traditional case-control study. Data from all first degree relatives of the glioma cases will be used in association studies and segregation analysis. In addition, we can screen DNA from members of multiplex families (families with 2 or more relatives with a primary CNS tumor) for mutations in candidate genes known to be associated with glioma, and contribute data from selected multiplex families to collaborative linkage studies to search for new genes conferring susceptibility to brain and possibly related tumors.

DETAILED DESCRIPTION:
To advance understanding of environmental, behavioral and genetic causes of brain tumors in adults, DCEG investigators initiated a multicenter case-control study of malignant and benign tumors in adults in 1994. This four-year study was conducted at participating hospitals in Boston, Phoenix, and Pittsburgh. Eligible cases were individuals greater than or equal to 18 years newly diagnosed with an intracranial glioma, meningioma or acoustic neuroma and treated at one of the participating hospitals. The controls were patients admitted to neurological, neurosurgical or general surgical services at the same three hospitals for any of a variety of non-neoplastic conditions. By the end of the study, 811 brain tumor cases had been accrued.

Information about a broad range of possible environmental, lifestyle, and genetic risk factors was obtained from both cases and controls through a computer-assisted personal interview (CAPI). The family history component obtained history and age at diagnosis of cancer or benign brain tumors and selected other diseases, for all living and deceased first degree relatives. A supplemental self-administered questionnaire covered diet, vitamin supplements, alcohol consumption, and household use of electrical appliances. Blood samples were obtained as a source of DNA. Currently, data analysis is in the early stages.

To increase our ability to examine both genetic and environmental components of brain tumor risk, we decided to add a family studies component to the case-control study, focusing on families of glioma cases. Initial contact with each family is made through the cases or, if a case is deceased, through the next of kin. Cases or next of kin are asked to complete a Family Health Questionnaire that updates the family medical history and provides contacting information for all adult first degree relatives and more distant relatives with cancer. Then, we contact all first degree relatives greater than or equal to age 18 years, and the next of kin of deceased eligible relatives and invite them to complete a modified risk factor interview conducted over the telephone. This interview obtains information about each relative s personal and family history of cancer and other diseases, and history of risk factor exposures, including all the major categories covered in the case-control study. Study participants who complete the interview are then asked to provide buccal cells as a source of DNA for future genotyping.

The glioma cases and their relatives will serve as a unique resource for both epidemiologic and genetic analyses. Selected relatives can serve as controls for association thereby eliminating concerns and population stratification. The study design also permits assessment of specific genetic hypotheses that cannot be evaluated in a traditional case-control study. Data from all first degree relatives of the glioma cases will be used in association studies and segregation analysis. In addition, we can screen DNA from members of multiplex families (families with 2 or more relatives with a primary CNS tumor) for mutations in candidate genes known to be associated with glioma, and contribute data from selected multiplex families to collaborative linkage studies to search for new genes conferring susceptibility to brain and possibly related tumors.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals who are eligible for this study include:

The 499 glioma cases who were interviewed for the case-control study between September, 1994 and July, 1998. The cases were enrolled through Joseph's Hospital and Medical Center (including Barrow Neurological Institute), Phoenix, AZ; Brigham and Women's Hospital, Boston, MA; and Western Pennsylvania Hospital, Pittsburgh, PA.

The following relatives greater than or equal to 18 years of age from simplex families: all first degree relatives; the spouse(s) of a case, if the spouse(s) had children with the case who are participating in the study.

The following relatives greater than or equal to 18 years of age from multiplex families: all first and second degree relatives; more distant blood relatives with cancer (secondary case); first degree relatives of every secondary case; the spouse(s) of every case or secondary case if the spouse(s) had children with the case or secondary case who are participating in the study; any blood relative not included above who connects a secondary case to a case.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: First-degree relatives of cases with malignant and benign brain tumors from a multi-center case-control study.
Sampling Method: Non-Probability Sample
Enrollment: 1871 (Actual)
Dates: Start 1999-03-11 (Actual); Primary Completion 2001-09-30 (Actual); Study Completion 2020-12-03 (Actual)

PRIMARY OUTCOMES:
Assess the roles of genetic susceptibility and environmental exposures in the risk of gliomas and related tumors | Underway
  Genetic susceptibility genes

CONTACTS AND LOCATIONS:
Overall Officials: Alisa M Goldstein, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - University of Arizona, Tucson, Arizona
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Western Pennsylvania Cancer Institute, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Inskip PD, Linet MS, Heineman EF. Etiology of brain tumors in adults. Epidemiol Rev. 1995;17(2):382-414. doi: 10.1093/oxfordjournals.epirev.a036200. No abstract available. PMID 8654518
- [Background] Halperin EC. Malignant gliomas in older adults with poor prognostic signs. Getting nowhere, and taking a long time to do it. Oncology (Williston Park). 1995 Mar;9(3):229-34; discussion 237-8, 243. PMID 7669516
- [Background] Greig NH, Ries LG, Yancik R, Rapoport SI. Increasing annual incidence of primary malignant brain tumors in the elderly. J Natl Cancer Inst. 1990 Oct 17;82(20):1621-4. doi: 10.1093/jnci/82.20.1621. PMID 2213902